CLINICAL TRIAL: NCT04366089
Title: Oxygen-Ozone as Adjuvant Treatment in Early Control of Disease Progression in Patients With COVID-19 Associated With Modulation of the Gut Microbial Flora
Brief Title: Oxygen-Ozone as Adjuvant Treatment in Early Control of COVID-19 Progression and Modulation of the Gut Microbial Flora
Acronym: PROBIOZOVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roberto Poscia MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Roberto Poscia MD, PhD, Medical Doctor, Azienda Policlinico Umberto I
Organization: Azienda Policlinico Umberto I (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110/2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID; SARS-CoV 2; Pneumonia, Viral; Coronavirus Infection
Keywords: Oxygen-ozone therapy; gut microbiota
MeSH Terms: conditions — Pneumonia, Viral; Coronavirus Infections | interventions — Standard of Care; Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Azithromycin 500mg 1 cp / day (alternatively lopinavir/ritonavir cps 200/50 mg, 2 cps x 2 / day or darunavir 800 mg 1 cp / day + ritonavir 100 mg 1 cp / day or darunavir/cobicistat 800/150 mg 1 cp / day), plus hydroxychloroquine cp 200 mg, 1 cp x 2 / day.
  Interventions: Drug: Azithromycin; Drug: hydroxychloroquine
- Oxygen-ozone and probiotic (Experimental): Oxygen-ozone therapy, probiotic supplementation plus standard of care
  Oxygen-ozone therapy: systemic autohemotherapy (twice a day).
  Probiotic supplementation: SivoMixx 200 billion (six sachets twice a day).
  Interventions: Other: Oxygen-ozone therapy, probiotic supplementation and Standard of care; Dietary Supplement: SivoMixx (200 billion); Drug: Azithromycin; Drug: hydroxychloroquine

INTERVENTIONS:
Other: Oxygen-ozone therapy, probiotic supplementation and Standard of care — - systemic autohemotherapy with Ozone 30 mcg / ml 250ml 2 times / day for 7 days
  Arms: Oxygen-ozone and probiotic
Dietary Supplement: SivoMixx (200 billion) — Composition of SivoMixx: Streptococcus thermophilus DSM322245, Bifidobacterium lactis DSM 32246, Bifidobacterium lactis DSM 32247, Lactobacillus acidophilus DSM 32241, Lactobacillus helveticus DSM 32242, Lactobacillus paracasei DSM 32243, Lactobacillus plantarum DSM 32244, Lactobacillus brevis DSM 27961 (NB: DSM n°... : bacterial strain identification code)
  Arms: Oxygen-ozone and probiotic
Drug: Azithromycin — dose: 500mg 1 cp / day (alternatively lopinavir/ritonavir cps 200/50 mg, 2 cps x 2 / day or darunavir 800 mg 1 cp / day + ritonavir 100 mg 1 cp / day or darunavir/cobicistat 800/150 mg 1 cp / day)
Drug: hydroxychloroquine — dose: 200 mg, 1 cp x 2 / day

SUMMARY:
Italy was the first European country affected by a severe outbreak of the Severe Acute Respiratory Syndrome - CoronaVirus-2 (SARS-CoV-2) epidemic emerged from Wuhan region (China), with a high morbidity and mortality associated with the disease.

In light of its pandemic spread and the very limited therapeutic options, COronaVIrus Disease 19 (COVID-19) is considered an unprecedented global health challenge. Therefore, the evaluation of new resources, designed in the first instance for other pathologies but potentially active against COVID-19, represents a priority in clinical research.

This is an interventional, non-pharmacological, open, randomized, prospective, non-profit study on the adjuvant use of oxygen ozone therapy plus probiotic supplementation in the early control of disease progression in patients with COVID-19.

Contextually, all patients are treated with the current standard of care on the basis of the interim guidelines of the Italian Society of Infectious and Tropical Diseases.

The main purpose of the study is to evaluate the effectiveness of an ozone therapy-based intervention (accompanied by supplementation with probiotics) in containing the progression of COVID-19 and in preventing the need for hospitalization in intensive care units.

DETAILED DESCRIPTION:
Several studies analyzed the mechanisms by which ozone therapy could combat viral infections. In particular, 1) the improvement of the release of oxygen in the peripheral tissues, 2) the anti-inflammatory action 3) a virucidal activity have been described.

In view of these properties, a number of international clinical trials on the topic are currently ongoing.

Hospitalization, dietary changes, use of antibiotics and systemic inflammation related to COVID-19 are all variables that contribute to changes in the intestinal and lung microbiota with significant repercussions on the outcomes of the disease. Furthermore, the use of ozone therapy could also lead to a modification of the microbial flora. Probiotic supplementation can help to correct these issues.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Nasopharyngeal swab positive for COVID-19
* COVID-19 stages I - II - III (*1)
* Hospitalization in the Department of Infectious Diseases

Exclusion Criteria:

* COVID-19 stages IV - V - VI (*1)
* Hospitalization in Intensive Care Units
* Pregnancy
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients who deny consent to the proposed treatment
* Inability to provide informed consent
* Contraindications to performing oxygen-ozone therapy
* hyperhomocysteinemia
* favism or thyroiditis
* coagulopathies
* neurodegenerative diseases
* angina (in particular Prinzmetal's angina) or with previous myocardial infarction

(*1) Compliant with indications published by:

Italian Society of Anesthesia Analgesia Resuscitation and Intensive Care (SIAARTI).

Care pathway for the patient with COVID-19.

Section 2 - Recommendations for local management of the critically ill patient - Version 2

Available on http://www.siaarti.it/SiteAssets/News/COVID19%20-%20documenti%20SIAARTI/Percorso%20COVID-19%20-%20Sezione%202%20-%20Raccomandazioni%20per%20la%20gestione%20locale%20-%20Rev%202.0.pdf

Last accessed 20/04/2020

Posted on 26.03.2020

On page 2 of the previous document :

"6 identified stages:

* sick disease - mild COVID-19 (I stage)
* light pneumonia - mild COVID-19 (II stage)
* serious pneumonia - severe COVID-19 (III stage)
* Acute respiratory distress syndrome (ARDS) - critical COVID-19 (IV stage)
* sepsis - critical COVID-19 (V stage)
* septic shock - critical COVID-19 (VI stage)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Delta in the number of patients requiring orotracheal intubation despite treatment | 21 days
  Comparison between the two groups

SECONDARY OUTCOMES:
Delta of crude mortality | 21 days
  Comparison between the two groups
Delta of length of stay for patients in hospital | 90 days
  Comparison between the two groups
delta in the value of interleukin (IL)-1 | 21 days
  Comparison between the two groups
delta in the value of IL-6 | 21 days
  Comparison between the two groups
delta in the value of IL-10 | 21 days
  Comparison between the two groups
delta in the value of Tumor Necrosis Factor (TNF)-alpha | 21 days
  Comparison between the two groups
delta in the value of cluster of differentiation (CD)4+ CD38/ Human Leukocyte Antigen-DR isotype (HLA-DR) | 21 days
  Comparison between the two groups
delta in the value of CD8+ CD38/ HLA-DR | 21 days
  Comparison between the two groups
delta in the value of fecal calprotectin | 21 days
  Comparison between the two groups
delta in the value of lipopolysaccharide (LPS) | 21 days
  Comparison between the two groups
delta in the value of zonulin | 21 days
  Comparison between the two groups
delta in the value of alpha1-antitrypsin | 21 days
  Comparison between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pugliese, MD, PhD, Principal Investigator — University of Rome Sapienza - Policlinico Umberto I Rome (Italy)
Locations (1):
- Francesco Pugliese, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hernandez A, Papadakos PJ, Torres A, Gonzalez DA, Vives M, Ferrando C, Baeza J. Two known therapies could be useful as adjuvant therapy in critical patients infected by COVID-19. Rev Esp Anestesiol Reanim (Engl Ed). 2020 May;67(5):245-252. doi: 10.1016/j.redar.2020.03.004. Epub 2020 Apr 14. PMID 32303365
- [Result] Conti P, Gallenga CE, Tete G, Caraffa A, Ronconi G, Younes A, Toniato E, Ross R, Kritas SK. How to reduce the likelihood of coronavirus-19 (CoV-19 or SARS-CoV-2) infection and lung inflammation mediated by IL-1. J Biol Regul Homeost Agents. 2020 March-April,;34(2):333-338. doi: 10.23812/Editorial-Conti-2. PMID 32228825
- [Result] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- See also: Clinical study for ozonated autohemotherapy in the treatment of Novel Coronavirus Pneumonia (COVID-19) — http://www.chictr.org.cn/showproj.aspx?proj=49947
- See also: A randomized controlled trial for the efficacy of ozonated autohemotherapy in the treatment of Novel Coronavirus Pneumonia (COVID-19) — http://www.chictr.org.cn/showproj.aspx?proj=49737
- See also: A multicenter randomized controlled trial for ozone autohemotherapy in the treatment of novel coronavirus pneumonia (COVID-19) — http://www.chictr.org.cn/showproj.aspx?proj=49747